CLINICAL TRIAL: NCT00854880
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Comparative Phase II Clinical Trial to Evaluate the Efficacy and Safety of PDC-339 for the Treatment of Acute Erosive Gastritis
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of PDC-339 for the Treatment of Acute Erosive Gastritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 921105; DOH94-TD-I-111-003
Record Dates: First submitted 2005-09-12; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2005-03

CONDITIONS: Erosive Gastritis
Keywords: Erosive Gastritis

INTERVENTIONS:
Drug: PDC339
Drug: Placebo

SUMMARY:
The objective of this trial is to evaluate the efficacy and safety of PDC-339 in the treatment of acute erosive gastritis, using placebo as the comparator.

DETAILED DESCRIPTION:
The primary biologically active components of ginseng are saponin triterpenoid glycosides called ginsenosides whose names relate to their chromatographic position (Ra, Rb, etc.). Based on the related studies, American ginseng was inferred to have the effects of modulating gastrointestinal system, lowering blood sugar level, enhancing memory, and suppressing mutation of breast cancer cell line. It also has anti-oxidant and neuroprotective effect. Among the experiences about the therapeutic uses of American ginseng, it is concluded that American ginseng is effective in treating gastrointestinal diseases. PDC339 is an active ingredient of American ginseng. This is a randomized, double blind, placebo-controlled parallel comparative phase II clinical trial to evaluate the efficacy and safety of PDC-339 in patients with acute erosive gastritis. The study period for each patient includes a screening/wash-out period of 1 week and a treatment period (including a 2-week follow-up) of 6 weeks. Subjects will be required to make a total of 5 visits. There will be a total of evaluable 60 patients (20 patients in each treatment group). If the drop out rate is assumed to be up to 10%, then there will be a total of 69 eligible patients. All of the subjects who meet the inclusion and exclusion criteria will be enrolled into the study and receive randomly either PDC-339 or placebo according a randomization list. The following clinical assessments will be performed: Primary efficacy assessment - the change of endoscopic gastric integrity; secondary efficacy assessment - the change of the severity of symptom on a 4-point scale at visit 3,4 from the baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 20 years old, male or female;
2. Patients have endoscopy-based evidence (Lanza Score ≧ 2) of untreated acute erosive gastritis at examination;
3. Having a negative result on a fecal occult blood test or hemoglobin below normal range of 2 g/dL;
4. Patients who voluntarily signed written informed consent may participate in the study.

Exclusion Criteria:

1. Pregnant or lactating female;*
2. Patients have endoscopy-based evidence of gastric malignancy, pyloric obstruction, and esophageal stricture requiring dilation, fresh clot, active bleeding, or perforated ulcers;
3. Use of any proton pump inhibitor, sucralfate, H2-receptor antagonist, or bismuth preparations within 1 week before initiating study drug therapy;
4. Patients requiring anticoagulants or corticosteroid therapy (at dosages greater than the equivalent of prednisone, 10 mg/day);
5. Patients with significant impairment of renal function (creatinine>2mg/dl); liver function impairment (AST and ALT 2x upper limit of normal); severe cardiac disease, e.g. angina pectoris, myocardial infarction, cardiac arrhythmia, congestive heart failure (New York Heart Association Functional Classification III and IV) or acute respiratory disease;
6. Any peptic ulcer at upper-gastrointestinal endoscopy;
7. Patients with a history of esophageal and/or gastric varices;
8. Known hypersensitivity to American ginseng;
9. Use of other investigational drugs within 30 days prior to the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
efficacy and safety of PDC-339

SECONDARY OUTCOMES:
improvement of clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D., Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan